CLINICAL TRIAL: NCT03852628
Title: Kappa Opioid Receptor Antagonism for the Treatment of Alcohol Use Disorder (AUD) and Comorbid Post-Traumatic Stress Disorder (PTSD)
Brief Title: Kappa Opioid Receptor Antagonism for the Tx of AUD and Comorbid PTSD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility analysis
Sponsor: Pharmacotherapies for Alcohol and Substance Use Disorders Alliance (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AS140026-A5
Record Dates: First submitted 2019-02-12; First posted 2019-02-25 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-04

CONDITIONS: Post Traumatic Stress Disorder; Alcohol Abuse
Keywords: Alcohol Use Disorder (AUD); Alcoholism; Alcohol Abuse; Post Traumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Buprenorphine; vivitrol

STUDY DESIGN:
Intervention Model Description: proof-of-concept study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To minimize bias, a placebo drug is employed as the comparison group to active study drug and the study is conducted in a double-masked fashion in that both the participants and the Independent Assessors who are assessing study outcomes are masked to treatment assignment. The only individuals at the site with access to treatment assignment information are the research pharmacists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2mg Buprenex and 380mg Vivitrol (Active Comparator): 2mg Buprenex and 380mg Vivitrol
  Buprenex (buprenorphine) 2mg sublingual (SL) (taken every day for 12 weeks) , with Vivitrol (naltrexone) 380mg intramuscular injection (IM) (given every 4 weeks)
  Interventions: Drug: 2mg Buprenex and 380mg Vivitrol
- Placebo (Placebo Comparator): Placebo (SL pill qd, IM injection q4weeks)
  Placebo pill (taken sublingual every day for 12 weeks) and IM placebo (given intramuscular injection, every 4 weeks at baseline, week4 and week8)
  Interventions: Drug: Placebo (SL pill qd, IM injection q4weeks)

INTERVENTIONS:
Drug: 2mg Buprenex and 380mg Vivitrol — Daily 2mg SL BUP (84 pills total, taken sublingual every day for 12 weeks) and Q4wks (given intramuscular, 3 injections total: at baseline, week4 and week8 ) IM NLTRX
  Other Names: 2mg Buprenex (SL, qd) and 380mg Vivitrol (IM, q4weeks); 2mg BUP/NLTRX
  Arms: 2mg Buprenex and 380mg Vivitrol
Drug: Placebo (SL pill qd, IM injection q4weeks) — Daily SL placebo (84 pills total, taken sublingual every day for 12 weeks) and Q4wks (given intramuscular, 3 injections total: at baseline, week4 and week8) IM Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Objective: Evaluate the efficacy and physiological effects of sublingual buprenorphine (SL-BUP; Subutex) combined with extended-release injectable naltrexone (XR-NTX; Vivitrol) in the treatment alcohol use disorder of comorbid (AUD) and post-traumatic stress disorder (PTSD)

DETAILED DESCRIPTION:
Hypothesis: The treatment of (sublingual buprenorphine) SL-BUP + (extended release naltrexone) XR-NTX will significantly reduce both (alcohol use disorder) AUD and (post-traumatic stress disorder) PTSD symptoms.

Primary Inclusion Criteria: Treatment-seeking individuals with comorbid AUD and PTSD

Subject Completion Target: A total of 90 male and female, treatment-seeking individuals with comorbid AUD and PTSD screened, enrolled, and randomized to treatment group

Study Protocol:

Screening: Potential participants are pre-screened by phone to ensure they meet basic study criteria. During informed consent and screening processes, participants receive thorough pre-enrollment education and the commitment to and feasibility for follow-up are confirmed. Screening visit is separate (at least 2-day interval) from Baseline visit. A participant who is otherwise meeting eligibility criteria except for taking an excluded medication can undergo a medically supervised discontinuation and 5-day washout of medication(s). At any point in the screening process and based on the inclusion and exclusion criteria listed above, the participant may be deemed eligible and proceed to baseline visit or investigator may exclude a participant and refer him/her for appropriate treatment.

At baseline, participants are randomized to receive either treatment A (buprenorphine 2mg SL with naltrexone 380mg IM) or treatment B (SL placebo and IM placebo) in a double-blind fashion. The treatment allocation ratio for the treatment vs. placebo regimens is 1:1.

At Screening, Baseline and Follow-up, an independent rater at each site performs the Timeline Follow Back (TLFB), Clinician Administered PTSD Scale for DSM-5 (CAPS-5), and Columbia Suicide Severity Rating (CSSR) assessments. Safety endpoints, adverse events (AEs), vital signs, and laboratory measures are tracked for each subject to assess study drug safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 70 years of age, capable of reading and understanding English, and able to provide written informed consent (i.e. no surrogate).
2. Current moderate to severe AUD as determined by MINI International Neuropsychiatric Interview for DSM-5 (MINI-5).
3. At least two recent episodes of heavy drinking (>5 standard drinks/sessions for men and >4 standard drinks/sessions for women) over the past 30 days, and heavy drinking pattern defined as 14 drinks per week for women and 21 drinks per week for men for at least 2 of a 4-week interval within the 90 days prior to baseline; i.e. at least Moderate Risk level on WHO category.
4. PTSD diagnosis defined by MINI-5 at screening.
5. Clinician Administered PTSD Scale for DSM-5 (CAPS-5) total score ≥26 for the past week at baseline.
6. Females of child-bearing potential must be using medically acceptable birth control (e.g. oral, implantable, injectable, or transdermal contraceptives; intrauterine device; double-barrier method) AND not be pregnant OR have plans for pregnancy or breastfeeding during the study.
7. Must have a CIWA-Ar score of < 8 prior to randomization.
8. Willing and able to refrain from medications thought to influence alcohol consumption (other formulations of naltrexone, disulfiram, acamprosate, topiramate, ondansetron, and baclofen).
9. Willing and able to refrain from psychotropic medications: stimulants/ADHD treatment, Alzheimer's medications, antipsychotics, benzodiazepines, antianxiety medications, mood stabilizers, and other sedatives.

   * Notes:

     * Participants may continue stable dose of antidepressants, prazosin, and non-benzodiazepine hypnotics and non-benzodiazepine anxiolytics to treat PTSD or insomnia.
     * Stable dose is defined as taken for ≥2 months prior to randomization and current does has been stable for ≥3 weeks prior to randomization and held constant during 12 weeks of study medication.)

Exclusion Criteria:

1. Current diagnosis of DSM-5 bipolar I, schizophrenia, schizoaffective, and/or major depressive disorder with psychotic features (defined by MINI-5 at screening).
2. Increased risk of suicide that necessitates inpatient treatment or warrants therapy excluded by the protocol, and/or current suicidal plan, per investigator clinical judgement, based on interview and defined on the Columbia Suicidality Severity Rating Scale (C-SSRS).
3. Treatment with trauma-focused therapy for PTSD (e.g. Cognitive Processing Therapy, Prolonged Exposure, or EMDR) within two weeks of baseline study visit. Note: Supportive psychotherapy in process for PTSD at time of Screening may be continued.
4. Current diagnosis of severe non-alcohol substance use disorder (except for caffeine and nicotine) during the preceding 1 month, based on participant screening interview.
5. Use of opioids within 2 weeks of baseline or opioid use disorder in the previous 90 days.
6. History of severe traumatic brain injury (TBI) per Ohio State University TBI Identification Method. Note: history of mild or moderate TBI is allowed.
7. Any clinically significant, uncontrolled, or medical/surgical condition that would contraindicate use of SL-BUP + XR-NTX, or limit ability to complete study assessments, including seizures (other than childhood febrile seizures), severe renal insufficiency, significant arrhythmia or heart block, heart failure, or myocardial infarction within the past 2 years, severe thrombocytopenia or hemophilia, severe hepatic failure, complete hearing loss, and/or need for surgery that might interfere with ability to participate.
8. Clinically significant laboratory abnormalities, including a thyroid stimulating hormone (TSH) >1.5 times upper limit of normal, hyperthyroidism, and aspartate aminotransferase and/or alanine aminotransferase > 3 times upper limit of normal; cardiovascular findings QTcF >500 msec on electrocardiogram (ECG) or blood pressure >190/110.
9. History of allergic reaction, bronchospasm or hypersensitivity to a naltrexone or buprenorphine.
10. Unable or unwilling to refrain from medications thought to influence alcohol consumption (see inclusion criteria above.)
11. Unable or unwilling to refrain from psychotropic medications (see inclusion criteria above); with the exception of stable doses of antidepressants, prazosin, and non-benzodiazepine hypnotics and non-benzodiazepine anxiolytics to treat PTSD or insomnia.
12. Persons who are imprisoned, of minor age, diagnosed with dementia, diagnosed with a terminal illness, or otherwise require a surrogate to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Davis, Principal Investigator — Associate Chief of Staff, Research & Development Service VA Medical Center
Locations (2):
- United States (2):
  - Tuscaloosa VA Medical Center, Tuscaloosa, Alabama
  - VA Connecticut Healthcare System, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
CDMRP has a policy to share and make available to the public the results and accomplishments of the activities that it funds. The PASA consortium plans to share de-identified data after final publication in a government-supported data repository.
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Groups:
- 2mg Buprenex and 380mg Vivitrol: 2mg Buprenex and 380mg Vivitrol
  Buprenex (buprenorphine) 2mg sublingual (SL) (taken every day for 12 weeks) , with Vivitrol (naltrexone) 380mg intramuscular injection (IM) (given every 4 weeks)
  2mg Buprenex and 380mg Vivitrol: Daily 2mg SL BUP (84 pills total, taken sublingual every day for 12 weeks) and Q4wks (given intramuscular, 3 injections total: at baseline, week4 and week8 ) IM NLTRX
- Placebo: Placebo (SL pill qd, IM injection q4weeks)
  Placebo pill (taken sublingual every day for 12 weeks) and IM placebo (given intramuscular injection, every 4 weeks at baseline, week4 and week8)
  Placebo (SL pill qd, IM injection q4weeks): Daily SL placebo (84 pills total, taken sublingual every day for 12 weeks) and Q4wks (given intramuscular, 3 injections total: at baseline, week4 and week8) IM Placebo
Period: Overall Study
Arm/Group | 2mg Buprenex and 380mg Vivitrol | Placebo
Started | 35 | 34
Completed | 22 | 22
Not Completed | 13 | 12
Not completed — Lost to Follow-up | 7 | 6
Not completed — Lack of Efficacy | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2mg Buprenex and 380mg Vivitrol | Placebo | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.9 (10.6) | 49.2 (13.1) | 50.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 29 | 28 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 20 | 38
  White | 13 | 13 | 26
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 3
Served in U.S. Military? [Count of Participants; unit: Participants] | 31 | 28 | 59
Anti-Depressant Use? [Count of Participants; unit: Participants] | 19 | 17 | 36
Enrolling Study Site [Count of Participants; unit: Participants]
  Tuscaloosa | 24 | 23 | 47
  West Haven | 11 | 10 | 21
  Wayne State University | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in Alcohol Use Disorder (AUD), With TLFB Tool
Description: Timeline Follow Back (TLFB) is a calendar-based method of assessing drinking patterns used to document the frequency and amount of daily alcohol consumption and to categorize the World Health Organization Risk Levels of Alcohol Use. An AUD reduction is defined as a WHO risk reduction of at least one category from baseline to week 8. The are 4 different WHO Risk Levels based on the grams of alcohol consumed per day: Very High Risk, High Risk, Medium Risk, and Low Risk (including abstinence).
Time Frame: Baseline and 8 weeks
Population: Includes all randomized participants that completed the baseline and Week 8 visit, and reported enough consecutive days of alcohol consumption at the week 8 visit (defined as being within one standard deviation of the population mean for the 28-day look back period).
Measure: Count of Participants; unit: Participants
Arm/Group | 2mg Buprenex and 380mg Vivitrol | Placebo
Number analyzed (Participants) | 30 | 28
Participants | 17 | 23
Statistical Analysis 1: Comparison: 2mg Buprenex and 380mg Vivitrol vs Placebo; The Placebo arm served as the reference group; Test type: Superiority; p = 0.08, Mixed Models Analysis; Modeled the probability of having a reduction in AUD; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.02 to 1.22]

2. Primary Outcome: Number of Participants With a Reduction in CAPS-5 Total Symptom Severity Score (TSSS) of 10 or More Points
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a 30-item structured interview to assess PTSD diagnosis and symptom severity. The CAPS-5 produces a PTSD Total Symptom Severity Score (TSSS) that ranges from 0 to 80, with a higher score indication worse PTSD symptoms. For this study, a reduction in PTSD symptoms is defined as a 10 or more point decrease in the CAPS-5 Total Symptom Severity Score (TSSS) from baseline to week 8.
Time Frame: Baseline and 8 weeks
Population: All randomized participants that completed the baseline and week 8 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | 2mg Buprenex and 380mg Vivitrol | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 14 | 15
Statistical Analysis 1: Comparison: 2mg Buprenex and 380mg Vivitrol vs Placebo; The placebo arm served as the reference group; Test type: Superiority; p = 0.690, Mixed Models Analysis; Modeled the probability of reduction in PTSD symptom; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.20 to 2.97]

3. Primary Outcome: Composite Outcome Measure for a Reduction in Both Alcohol Use Disorder (AUD) and Post-Traumatic Stress Disorder (PTSD) Symptoms
Description: AUD is measured by the Timeline Follow Back (TLFB). This instrument documents the amount of daily alcohol consumption (in grams) and categorizes the World Health Organization Risk Levels of Alcohol Use. The are 4 different WHO Risk Levels: Very High Risk, High Risk, Medium Risk, and Low Risk (including abstinence). An AUD reduction is defined as a WHO risk reduction of at least one category from baseline to week 8. PTSD symptom is measured by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). This 30-item interview assesses PTSD diagnosis and symptom severity. The CAPS-5 Total Symptom Severity Score (TSSS) ranges from 0 to 80, with higher scores indicating worse symptoms. A reduction in PTSD symptom is defined as a 10+ point decrease in the TSSS from baseline to week 8. A positive response for the composite primary outcome measure is defined as at least a 1-category risk reduction on the WHO s and at least a 10-point decrease in TSSS from baseline to Week 8.
Time Frame: Baseline and 8 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 2mg Buprenex and 380mg Vivitrol | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 10 | 12
Statistical Analysis 1: Comparison: 2mg Buprenex and 380mg Vivitrol vs Placebo; The Placebo arm served as the reference group; Test type: Superiority; p = 0.52, Mixed Models Analysis; Modeled the probability of have both a reduction in PTSD and AUD; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.15 to 2.66]

ADVERSE EVENTS:
Time Frame: From baseline visit (after first treatment allocation) through the Week 14 study visit.
Arm/Group | 2mg Buprenex and 380mg Vivitrol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 3/35 | 0/34
Other Adverse Events (participants affected / at risk) | 22/35 | 16/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg Buprenex and 380mg Vivitrol (N=35) | Placebo (N=34)
Congestive Heart Failure, Exacerbation (Cardiac disorders) | 1 (1) | 0 (0)
Fractured Vertebrae (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg Buprenex and 380mg Vivitrol (N=35) | Placebo (N=34)
Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acid reflux (esophageal) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 (3) | 0 (0)
Alcoholic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety aggravated (Psychiatric disorders) | 1 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (3)
Chills (Gastrointestinal disorders) | 0 (0) | 2 (3)
Congestive cardiac failure aggravated (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crawling Sensation (Nervous system disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diastolic BP increased (Investigations) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (5)
Fibromyalgia worsened (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fractured vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Heart racing (Cardiac disorders) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 6 (7) | 5 (5)
Knee Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine aggravated (Nervous system disorders) | 0 (0) | 1 (1)
Myalgia of lower extremities (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Nightmares (Psychiatric disorders) | 0 (0) | 1 (1)
Numbness of tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
Product used for unknown indication (Surgical and medical procedures) | 0 (0) | 1 (1)
Pulse increased (Investigations) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Short-term memory loss (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Visual disturbances (Eye disorders) | 1 (1) | 0 (0)
Vivid dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weakness (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
There are no secondary outcome results to report as this study was closed for futility before enough data was collected to report secondary outcomes. .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03852628/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03852628/SAP_001.pdf
  • Informed Consent Form (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT03852628/ICF_002.pdf